CLINICAL TRIAL: NCT05798533
Title: The Neoantigen Targeting T Cells Suspension for Intravenous Infusion(Neo-T) in Treating Patients With Advanced Solid Tumor
Brief Title: Neo-T in Treating Patients With Advanced Solid Tumors(GI-NeoT-03)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BGI, China (Other)
Collaborators: Fudan University (Other); Shanghai 10th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGI-004
Record Dates: First submitted 2023-03-23; First posted 2023-04-04 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-03

CONDITIONS: Solid Tumor
Keywords: Melanoma; non-small cell lung cancer; NSCLC; Neoantigen; Adoptive T cell Therapy
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — Infusions, Intravenous; toripalimab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of Neo-T and anti-PD1 (Experimental): Dose escalation will use a 3+3 design and will enroll cohorts of 3-6 patients with MEL or NSCLC at escalating doses of 1.2×10^9 cells and 3.6×10^9 cells.
  Interventions: Biological: Neo-T; Combination Product: Toripalimab; Combination Product: Tislelizumab

INTERVENTIONS:
Biological: Neo-T — Patients will receive Neo-T iv on day 0. Three times of cell infusion with an interval of 7 days constitute a cycle,maximum four cycles of treatment for patients.
  Other Names: Neoantigen targeting T cells Suspension for Intravenous Infusion
Combination Product: Toripalimab — 3mg/kg iv; Within 7 days after the first PBMC collection (day-38±3), the first dose was administered, and thereafter every 2 weeks.
  Toripalimab is recommended for patients with Melanoma.
  Other Names: JS001
Combination Product: Tislelizumab — 200mg iv; Within 7 days after the first PBMC collection (day-38±3), the first dose was administered, and thereafter every 3 weeks.
  Tislelizumab is recommended for patients with NSCLC or other tumor types.
  Other Names: BGB-A317

SUMMARY:
The primary objective of this study is to evaluate the safety of Neo-T in combination with anti-PD1 in patients with solid tumors.

The secondary objective of this study is to evaluate preliminarily the effect of Neo-T in combination with anti-PD1 in patients with solid tumors.

DETAILED DESCRIPTION:
This is a single arm, open label and non-randomized clinical study.

6 to12 patients will be enrolled to assess the safety and explore recommended dose of Neo-T combined with anti-PD1.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than or equal to 18 years of age and less than or equal to 75 years of age; all genders.
2. Advanced solid tumors including but not limited to some high frequency somatic mutations,such as melanoma,driver mutation-negative non-small cell lung cancer.
3. Advanced solid tumors patients who are HLA - A0201 /A1101/A2402 subtypes.
4. Measurable solid tumors with at least one lesion that is resectable or tumor biopsies for DNA extraction.
5. Patients who failed or were intolerant to standard treatment.
6. Possess venous access for mononuclear cell collection or intravenous blood collection.
7. Patients (or their legal representatives) who are able to understand and sign the Informed Consent Form and willing to sign a durable power of attorney.
8. Clinical performance status of ECOG is 0 or 1.
9. Patients who are able to cooperate to observe adverse reactions and the effect of the treatment,expected lifetime is greater than six month.
10. Patients of both genders must be willing to practice birth control from the time of enrollment to three months after treatment on this study,a fertile woman must have a negative pregnancy test.
11. The laboratory test values and the functions of important organs meet the following requirements:1）Serology: HIV antibody(-), hepatitis B DNA(-), hepatitis C antibody(-) and no active syphilis infection; 2）Hematology: Absolute neutrophil count is greater than or equal to 1.5×10^9/L; WBC is greater than or equal to 3×10^9/L; lymphocyte count is greater than or equal to 0.8×10^9/L; Platelet count is greater than or equal to 80×10^9/L; Hemoglobin is greater than or equal to 90g/L ; 3）Chemistry: Serum ALT/AST is less than or equal to 3 times ULN,except in patients with liver metastasis who must have ALT/AST less than or equal to 5 times ULN; Serum Creatinine is less than or equal to 1.5 times ULN ; Total bilirubin is less than or equal to 1.5 times ULN, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 times ULN;4）Blood Clotting Parameters:Prothrombin Time(PT) and International Normalised Ratio (INR) are less than or equal to 1.5 times ULN;Activated Partial Thromboplastin Time (APTT) is less than or equal to 1.5 times ULN;For subjects who frequently take anticoagulant drugs,their blood clotting parameters can meet the value range adaptive to this special population;5）Left ventricular ejection fraction（LVEF）is more than or equal to 50%.
12. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the first dose of anti-PD1, and toxicities must have recovered to grade 1 or less (except for toxicities such as alopecia or vitiligo).

Exclusion Criteria:

1. Pregnant or lactating women.
2. History of severe immediate hypersensitivity reaction to Neo-T and any of the agents used in this study.
3. Subjects with a history of organ transplantation.
4. Subjects with brain metastases.
5. Any active autoimmune disease or subjects with a history of autoimmune diseases that have been assessed by the investigator to be unsuitable for this study.Including but not limited to the following diseases: such as systemic lupus erythematosus, immune related neuropathy, multiple sclerosis, Guillain Barre syndrome, myasthenia gravis, connective tissue diseases, inflammatory bowel diseases(Crohn's disease and ulcerative colitis), excluding vitiligo, eczema, type I diabetes, rheumatoid arthritis and other joint diseases, Sjogren's syndrome and controlled psoriasis by local medication.
6. Active systemic infections,for example, acute infections requiring systemic antibiotic, antiviral, or antifungal treatment occur within 2 weeks before enrollment.
7. Severe liver and kidney function damage(unable to control after treatment,and biochemical indicators cannot meet the Exclusion Criteria of 11th), uncontrollable diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease, or poorly controlled hypertension (systolic pressure>160mmHg and/or diastolic pressure>90mmHg); active cardiovascular and cerebrovascular diseases, such as acute stroke,myocardial infarction,unstable angina,congestive heart failure rated as Grade II or above by the New York Heart Association, severe cardiac arrhythmias that cannot be controlled with medication,electrocardiograms show significant abnormalities (three consecutive times with an interval of at least 5 minutes) which have been assessed by the investigator that affect subsequent cellular treatment; mental illness and drug abuse, or any situation that the investigator assessments may increase the risk of this study.
8. Subjects plan to receive glucocorticoid(the dose of prednisone or alternative drug is more than 10mg per day) or other immunosuppressant within 4 weeks before the first dose of anti-PD1.Tips: when there is no active autoimmune disease, it is allowed to use prednisone or alternative drug with a dose less than 10 mg per day; Allowing subjects to use topical, ocular, intra articular, intranasal, and inhaled glucocorticoids for treatment.
9. Subjects plan to receive immunomodulatory drugs (such as interferon, GM-CSF, thymosin, gamma globulin, excluding IL-2) within 4 weeks before the first dose of anti-PD1.
10. The investigator assessed that the subject was unable or unwilling to comply with the requirements of the study protocol.
11. The genes correlated to functional defects in antigen presentation, antigen recognition, and cell killing have been detected.
12. With a history of other malignant tumors within the past 5 years; Excluding basal cell carcinoma, thyroid papillary carcinoma, cervical carcinoma in situ, or breast ductal carcinoma in situ.
13. The subject has any disease or medical condition that may affect the safety or effectiveness evaluation of the study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v5.0. | one month
  Keep records the adverse events experienced by subjects in 28 days after the first infusion.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | one year
  ORR is defined as the proportion of participants with tumor size reduction(CR,PR) assessed by RECIST 1.1 and iRECIST.
Disease Control Rate(DCR) | one year
  DCR is defined as the proportion of participants with tumor size reduction(CR,PR) and stable disease(SD) assessed by RECIST 1.1 and iRECIST.
Overall survival(OS) | one year
  The time from the first infusion of Investigational Product until death.
Progression-free survival(PFS) | one year
  PFS is defined as the time from the first infusion of Investigational Product until objective tumor progression, as assessed by RECIST 1.1 and iRECIST, or death, whichever occurs first.
Duration of Response(DOR) | one year
  DOR refers to the period from the first evaluation of tumor as CR or PR to the first evaluation as PD(Progressive Disease) per RECIST1.1 and iRECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Doctor, Principal Investigator — Fudan University; Yong Chen, Doctor, Principal Investigator — Fudan University; Qing Xu, Doctor, Principal Investigator — Shanghai 10th People's Hospital
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li D, Chen C, Li J, Yue J, Ding Y, Wang H, Liang Z, Zhang L, Qiu S, Liu G, Gao Y, Huang Y, Li D, Zhang R, Liu W, Wen X, Li B, Zhang X, Zhang X, Xu RH. A pilot study of lymphodepletion intensity for peripheral blood mononuclear cell-derived neoantigen-specific CD8 + T cell therapy in patients with advanced solid tumors. Nat Commun. 2023 Jun 10;14(1):3447. doi: 10.1038/s41467-023-39225-7. PMID 37301885
- [Background] Guo Z, Yuan Y, Chen C, Lin J, Ma Q, Liu G, Gao Y, Huang Y, Chen L, Chen LZ, Huang YF, Wang H, Li B, Chen Y, Zhang X. Durable complete response to neoantigen-loaded dendritic-cell vaccine following anti-PD-1 therapy in metastatic gastric cancer. NPJ Precis Oncol. 2022 Jun 3;6(1):34. doi: 10.1038/s41698-022-00279-3. PMID 35661819